CLINICAL TRIAL: NCT06105476
Title: Effect of Protein and Retinol on Alcohol-induced FGF21
Acronym: FGF21-APA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: FGF21-APA
Record Dates: First submitted 2023-10-12; First posted 2023-10-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Healthy
MeSH Terms: interventions — Ethanol; Vitamin A

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Alcohol (Experimental)
  Interventions: Other: Alcohol
- Alcohol+protein (Experimental)
  Interventions: Other: Alcohol+protein
- Alcohol+retinol (Experimental)
  Interventions: Other: Alcohol+retinol
- Retinol (Experimental)
  Interventions: Other: Retinol

INTERVENTIONS:
Other: Alcohol — Test drink with 12 g alcohol (30 g vodka 40%) in water
  Arms: Alcohol
Other: Alcohol+protein — Test drink with 12 g alcohol (30 g vodka 40%) and 25 g whey protein in water
  Arms: Alcohol+protein
Other: Alcohol+retinol — Test drink with 12 g alcohol (30 g vodka 40%) and 1000 μg retinol in water
  Arms: Alcohol+retinol
Other: Retinol — Test drink with 1000 μg retinol in water
  Arms: Retinol

SUMMARY:
The aims of this study are two-fold. First to investigate the influence of protein on the FGF21 response induced by alcohol, and second to investigate the influence of retinol on FGF21 concentrations and the FGF21 response induced by alcohol. Exploratory, and in order to investigate mechanisms behind the potential influence on alcohol-induced FGF21 response from protein or retinol intake, plasma glucose, insulin, glucagon, ethanol, acetaldehyde, acetate, retinol, retinoic acid, as well as subjective rating of appetite, will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Healthy men and women
* Age between 18 and 50 years
* Body mass index (BMI) between 20 and 27 kg/m2

Exclusion Criteria:

* Chronic diseases or significant health problems that are disruptive for participation in the study (as judged by the principal investigator/clinical responsible)
* Use, currently or within the previous 3 months, of medication that has the potential of affecting any of the blood parameters assessed in the study (as judged by the investigators)
* Blood donation within the last 3 months or during the study period
* Regular smoking or other nicotine use (electronic cigarettes, gum, snus, etc.) or nicotine cessation within the past 3 months.
* Currently dieting or having lost/gained a significant amount of weight (±3 kg) in the previous 3 months
* Women who are pregnant, breast-feeding or have the intention of becoming pregnant during the study period
* Food allergies or food intolerance relevant for the study (judged by the investigators)
* Substance abuse (alcohol and/or drugs) within the last 12 months
* Average weekly alcohol intake above the recommendations from the Danish Health and Medicines Authority (10 standard units per week)
* Taking dietary supplements containing vitamin A during the past 3 months
* Simultaneous participation in other clinical studies that can interfere with the current study
* Inability, physically or mentally, to comply with the procedures required by the study protocol

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Plasma FGF21 response after consumption of alcohol+protein vs alcohol | Outcomes are measured at time 0, 30, 60, 120, 180, and 240 minutes after test drinks.
  Time*drink interaction and iAUC
Plasma FGF21 response after consumption of alcohol+retinol vs alcohol vs retinol | Outcomes are measured at time 0, 30, 60, 120, 180, and 240 minutes after test drinks.
  Time*drink interaction and iAUC

SECONDARY OUTCOMES:
Plasma glucose, insulin, glucagon, ethanol, acetaldehyde, acetate, retinol, and retinoic acid after consumption of alcohol+protein vs alcohol+retinol vs alcohol vs retinol. | Outcomes are measured at time 0, 30, 60, 120, 180, and 240 minutes after test drinks.
  Time*drink interaction and iAUC
Subjective appetite ratings after consumption of alcohol+protein vs alcohol+retinol vs alcohol vs retinol. | Outcomes are measured at time 0, 30, 60, 120, 180, and 240 minutes after test drinks.
  Time*drink interaction and iAUC

CONTACTS AND LOCATIONS:
Overall Officials: Niels Grarup, Principal Investigator — Novo Nordisk Foundation Center for Basic Metabolic Research, Health and Medical Sciences, University of Copenhagen
Locations (1):
- Departmen of Nutrition, Exercise and Sports, Copenhagen, Denmark